CLINICAL TRIAL: NCT05943756
Title: Evaluation of Well-being Interventions in Adults With TBI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kessler Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E-1220-23
Record Dates: First submitted 2023-07-05; First posted 2023-07-13 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: TBI (Traumatic Brain Injury)
Keywords: TBI, Traumatic Brain Injury, Traumatic Injury, Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Intervention Model Description: Both groups will participate in a different intervention program meant to improve well-being in individuals who have sustained a brain injury.
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Signature Strengths (Experimental): In this arm, participants would participate in in an intervention program meant to improve well-being in individuals who have sustained a brain injury.
  Interventions: Behavioral: Signature Strengths
- TBI Education Course (Active Comparator): In this arm, participants would participate in in an intervention program meant to improve well-being in individuals who have sustained a brain injury.
  Interventions: Behavioral: TBI Education Course

INTERVENTIONS:
Behavioral: Signature Strengths — The treatment group will complete 6 web-based sessions of Signature Strengths(1 sessions per week for 6 weeks), designed to teach lessons focused on the Aware-Explore-Apply interventional framework. Sessions are approximately 60 minutes long.
  Arms: Signature Strengths
Behavioral: TBI Education Course — The control group will complete 6 web-based sessions of a TBI Education Course(1 sessions per week for 6 weeks), designed to teach lessons based on the TBI Model Systems Knowledge Translation Center's fact sheets. Sessions are approximately 60 minutes long.
  Arms: TBI Education Course

SUMMARY:
The purpose of this research is to evaluate the potential benefits of two Intervention programs in adults with TBI to improve well-being and other outcomes that are maintained over time.

DETAILED DESCRIPTION:
The current study will examine the efficacy of Signature Strengths in adults with TBI to improve self-concept and other outcomes that are maintained over time. Preliminary evidence suggests that after a TBI, an individual can experience significant alteration to their personal identity and a perceived loss of their pre-injury self. By using this Signature Strength intervention, adults with moderate to severe TBI will be able to become aware of their most used "signature" strengths, explore how these strengths are used in everyday life, and apply them in future situations to bring well-being and to better cope with stressors.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Have a diagnosis with moderate to severe TBI
* At least one year post injury
* Able to speak and read English fluently

Exclusion Criteria:

* Have a history of multiple sclerosis, stroke, seizures or another nervous system injuries disease in the past (like brain tumor or epilepsy)
* Have a significant psychiatric illness (like, schizophrenia or psychosis)
* Currently taking steroids and/or benzodiazepines as determined by study staff review of medications
* Significant alcohol or drug abuse history (requiring inpatient treatment)
* History of stroke, schizoaffective disorder, bipolar disorder, personality disorder or severe depression determined by extensive screening by a trained staff member
* Previous participation in a Signature Strengths program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2023-09-25 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Rosenberg Self-Esteem Scale (RSES) | Baseline, 3 months posttest, and 6 months posttest
  Self-report self-esteem questionnaire. Values range from 10-40, with higher score indicating better outcome.
Strengths Knowledge and Strengths Use Scale (SKUS) | Baseline, 3 months posttest, and 6 months posttest
  Measure to assess knowledge and use of one's strengths and measure changes following strengths-based interventions. Two scores: Strengths Use and Strengths Knowledge. Strengths Use values range from 14-98, with higher score indicating a better outcome. Strengths Knowledge values range from 8-56, with higher score indicating a better outcome.
Head Injury Semantic Differential Scale - Version III (HISD-III) | Baseline, 3 months posttest, and 6 months posttest
  Self-report for examination of past and present self-identity. Values range from 18-126, with higher score indicating a better outcome.
Global Assessment of Character Strengths | Baseline, 3 months posttest, and 6 months posttest
  24-item questionnaire to rate levels of individual's character strengths. Values range from 24-120, with higher score indicating a better outcome.
Twenty-Statements Task | Baseline, 3 months posttest, and 6 months posttest
  20-item questionnaire used to measure an individual's self concept filling out the twenty items that each start with the words "I am..." which will be analyzed for positive and negative valence, with higher score indicating a better outcome. There is no maximum or minimum value for this test.

SECONDARY OUTCOMES:
Flourishing Scale (FS) | Baseline, 3 months posttest, and 6 months posttest
  Measure of well-being and "flourishing". Values range from 8-56, with higher score indicating a better outcome.
Quality of Life After Brain Injury (QOLIBRI) | Baseline, 3 months posttest, and 6 months posttest
  Assess Quality of Life specifically in Brain Injury. Values range from 0-100, with higher score indicating a better outcome.
Satisfaction with Life Scale (SWLS) | Baseline, 3 months posttest, and 6 months posttest
  Measure of life satisfaction. Values range from 5-35, with higher score indicating a better outcome.
Positive and Negative Affect Schedule (PANAS) | Baseline, 3 months posttest, and 6 months posttest
  Measure of both positive and negative emotional feelings. Values range from 10-50, with higher score indicating a better outcome.
Voicemail Elicitation Task | Baseline, 3 months posttest, and 6 months posttest
  Measures how individuals respond to social situations using politeness/impoliteness. Values are calculated by dividing the total number of politeness markers by the total time in minutes, with a higher score indicating a better outcome. There are no minimum or maximum values for this test.
Perceived Stress Scale | Baseline, 3 months posttest, and 6 months posttest
  10 item, Self-report measure of perceived stress. Values range from 0-40, with higher score indicating a worse outcome.
Connor-Davidson Resilience Scale 10 (CD-RISC-10) | Baseline, 3 months posttest, and 6 months posttest
  10 item self-report measure of resilience. Values range from 0-40, with higher score indicating a better outcome.
Brain Injury Self-Efficacy Scale | Baseline, 3 months posttest, and 6 months posttest
  20 item self-report measure of self-efficacy and coping. Values range from 0-80, with higher score indicating a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Helen Genova, Ph. D., Principal Investigator — Kessler Foundation
Locations (1):
- Kessler Foundation, East Hanover, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No